CLINICAL TRIAL: NCT05690698
Title: Quetiapine Versus Haloperidol in the Management of Hyperactive Delirium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QHMHD
Record Dates: First submitted 2022-12-28; First posted 2023-01-19 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-03

CONDITIONS: Hyperactive Delirium
Keywords: Critical Care; Hyperactive Delirium; antipsychotics; Haloperidol; Quetiapine
MeSH Terms: interventions — Haloperidol

STUDY DESIGN:
Intervention Model Description: Parallel random assignment to receive either oral quetiapine (25-50 mg/day) or haloperidol (1-2 mg/day)
Who Masked: Participant, Care Provider
Masking Description: Double blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quatiapine group (n=50) (Experimental): Quetiapine (25-50 mg/day) according to their symptoms of agitations.
  Interventions: Drug: Quatiapine
- Haloperidol group (n=50) (Active Comparator): Haloperidol (1-2 mg/day) according to their symptoms of agitations.
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Quatiapine — Atypical antipsychotic
  Arms: Quatiapine group (n=50)
Drug: Haloperidol — Antipsychotic
  Arms: Haloperidol group (n=50)

SUMMARY:
In population of intensive care unit (ICU), most studies compared atypical antipsychotics such as quetiapine with the traditional haloperidol in delirious patients of various forms and etiologies. The role of such agents in patients with hyperactive is not fully understood.

This study compares the effectiveness of quetiapine with haloperidol in treating the hyperactive form of delirium in terms of their effects on morbidity, length of stay in the intensive care unit, and mortality in critically ill patients.

DETAILED DESCRIPTION:
A common complication in the intensive care unit (ICU) that has recently been identified is delirium. Defining delirium as a "sudden deterioration in attention, awareness, and cognition, which is not explained by any pre-existing neurocognitive disorder, but because of another medical condition," the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) clarified the definition of delirium.

A dibenzothiazepine derivative with a novel and distinctive pharmacologic profile is quetiapine. The limbic system is overactive in delirium, which is one of its pathophysiologies. By obstructing the mesolimbic dopamine D2 receptors specifically, quetiapine may be able to regulate this hyperactivity.

The objective of this study is to compare the effectiveness of quetiapine with haloperidol in treating the hyperactive form of delirium in terms of their effects on morbidity, length of stay in ICU, and mortality in critically ill patients.

This research will not receive any grants, funding, or financial aid (NOT FUNDED STUDY). Collaborators declare that they have no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are diagnosed with hyperactive form of delirium during their ICU stay using CAM-ICU tool (the confusion assessment method for the intensive care unit)

Exclusion Criteria:

* Suspected substance-induced delirium
* Previous use of antipsychotics
* Known allergy or intolerance to the study drugs
* Pregnancy or breast feeding
* Acute renal injury
* Hepatic failure
* Inability to tolerate oral drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-04-09 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Response rate | Day 7
  Response rate is defined as a reduction of the DRS-R-98 severity score from its baseline for 50% or more and a DRS-R-98 severity score of 12 or less without relapse

SECONDARY OUTCOMES:
In-hospital mortality | week 6 from enrollment
  In-hospital all cause mortality
ICU-mortality | week 6 from enrollment
  ICU all cause mortality
Need for MV | week 6 from enrollment
  Need for mechanical ventilation during ICU stay
ICU stay | week 6 from enrollment
  Number of days of ICU stay
Hospital stay | week 6 from enrollment
  Number of days of hospital stay

OTHER OUTCOMES:
Sleeping hours | Day 3
  Sleeping hours per night
Sleeping hours | Day 7
  Sleeping hours per night
Delirium Rating Scale-revised-98 severity score | Day 3
  The DRS-R-98 is a valid measure of delirium severity over a broad range of symptoms and is a useful diagnostic and assessment tool, maximum severity score of 39 points
Delirium Rating Scale-revised-98 severity score | Day 7
  The DRS-R-98 is a valid measure of delirium severity over a broad range of symptoms and is a useful diagnostic and assessment tool, maximum severity score of 39 points

CONTACTS AND LOCATIONS:
Overall Officials: Tamer N. Habib, MD, Principal Investigator — University of Alexandria; Islam E. Ahmed, PharmD, Study Chair — Faculty of Medicine, Suez-canal University; Ibrahim K. Luttfi, PHD, Study Director — Faculty of Medicine, Gezira University
Locations (1):
- Faculty of Medicine, Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No